CLINICAL TRIAL: NCT05168579
Title: Developing a Deliberate Practice Intervention to Recalibrate Physician Heuristics in Trauma Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Deepika Mohan, Associate Professor of Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20120026; R21AG072072 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: two arm randomized trial
Who Masked: Outcomes Assessor
Masking Description: Allocation to treatment v. control group will be masked to the person doing the analysis until the data is locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deliberate practice (Experimental): Trainees will be paired with a coach, and will meet, once per week for thirty minutes, over a three week period. During the training session, coach-trainee dyads will play a puzzle video game, and will discuss contextual cues that should inform triage decisions. At the completion of the three weeks, trainees will complete a semi-structured, debriefing interview and a virtual simulation to assess triage performance.
  Interventions: Behavioral: Deliberate practice
- Control (No Intervention): Participants in the control group will complete a virtual simulation.

INTERVENTIONS:
Behavioral: Deliberate practice — As above
  Arms: Deliberate practice

SUMMARY:
The objective of this study is to test the feasibility of using deliberate practice - goal-oriented training in the presence of a coach who can provide personalized, immediate feedback - to increase engagement. The research design involves recruitment of a national convenience sample of board-certified emergency physicians who will serve as trainees (n=30), pairing of the trainees with a coach, delivery of three 30-minute coaching sessions using the existing games as the training task, and assessment of the effect of the combined intervention on performance in the laboratory. The specific aims are:

1. To assess the fidelity of intervention delivery by measuring coaching skill acquisition, coaching skill drift and protocol adherence.
2. To assess the potential effect size of the intervention by comparing trainee performance on a validated virtual simulation with a control group of physicians (n=30).
3. To assess the acceptability of the intervention by using a mixture of validated instruments and semi-structured debriefing interviews with trainees to assess their engagement with the intervention.

DETAILED DESCRIPTION:
Deliberate practice - goal-oriented training in the presence of a coach who can provide personalized, immediate feedback - has successfully improved performance across multiple domains, including sports, music, and combat. When used in conjunction with simulation to improve surgical skill, it has a large effect on educational outcomes. It has characteristics that make its application in this context potentially powerful (e.g. personalized feedback/relationship with coach increase engagement) but also potentially challenging (e.g. the diagnostic process does not lend itself easily to assessment). The objective of this study is to test the feasibility of using deliberate practice to amplify the effect of a video game intervention. The team will recruit a national sample of board-certified emergency physicians (n=30) to serve as trainees, with members of the team (n=3) serving as coaches. Trainee-coach dyads will meet for 30 minutes/week for 3 weeks, by video-conferencing, to play one of the existing video games and to use it to practice pattern recognition. Aims are:

1. To assess the fidelity of intervention delivery. Approach: the team will standardize coaching skill during an 'on-boarding session,' measure skill drift over the course of training sessions, and measure protocol adherence (primary outcome). Hypothesis: >90% of dyads will complete three training sessions.
2. To assess the potential effect size of the intervention. Approach: the team will compare performance of trainees (n=30) with a control group of physicians (n=30) on a validated virtual simulation. Hypothesis: Trainees will make ≥25% fewer diagnostic errors than control physicians (large effect size).
3. To assess the acceptability of the intervention. Approach: the team will conduct semi-structured debriefing interviews with trainees, assessing elements of the intervention that promote engagement.

This proposal will inform a future Stage III trial to compare the effect of different interventions on diagnostic error in trauma triage. If successful, this program of research will have an impact on patients by reducing the burden imposed by injury and by addressing the refractory problem of diagnostic error. It is novel conceptually in its effort to make heuristics a source of power, methodologically in its use of deliberate practice to improve diagnosis, and translationally in its use of video game technology. It is feasible because the investigative team has clinical and behavioral science expertise, experience developing deliberate practice interventions, and a track record of successfully building video games that can transform physician behavior. It responds to two national research priorities: 1) improving the diagnostic process; 2) maintaining health and independent living among the aging.

ELIGIBILITY:
Inclusion Criteria:

Board certified physicians who work at non-trauma centers in the United States

Exclusion Criteria:

Physicians without board certification (i.e., residents). Physicians who work only at trauma centers in the US.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Mohan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared with researchers conditional on approval from the University of Pittsburgh Office of Research
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available at the conclusion of the analytic phase of the trial, and for 3 years thereafter.
Access Criteria: Access will be provided to researchers and interested parties.

REFERENCES:
- [Derived] Mohan D, Elmer J, Arnold RM, Forsythe RM, Fischhoff B, Rak K, Barnes JL, White DB. Testing a Novel Deliberate Practice Intervention to Improve Diagnostic Reasoning in Trauma Triage: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2313569. doi: 10.1001/jamanetworkopen.2023.13569. PMID 37195666
- [Derived] Mohan D, Elmer J, Arnold RM, Forsythe RM, Fischhoff B, Rak K, Barnes JL, White DB. Testing the feasibility, acceptability, and preliminary effect of a novel deliberate practice intervention to reduce diagnostic error in trauma triage: a study protocol for a randomized pilot trial. Pilot Feasibility Stud. 2022 Dec 12;8(1):253. doi: 10.1186/s40814-022-01212-y. PMID 36510328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single email invitation was sent to 633 physicians who had previously participated in research (with valid contact information), asking them to forward the invitation to two colleagues. 78 responses were received. Five were excluded because they lived outside the contiguous 48 US States (e.g., in Canada or Puerto Rico) and one was excluded for refusing to consent to videotaping.
Period: Overall Study
Arm/Group | Deliberate Practice | Control
Started | 36 | 36
Completed | 30 | 21
Not Completed | 6 | 15
Not completed — Lack of Consent | 1 | 0
Not completed — Conflicts with time | 2 | 0
Not completed — Time slots were full | 3 | 0
Not completed — Lost to Follow-up | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deliberate Practice | Control | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 35 | 33 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast | 10 | 9 | 19
  United States: Southeast | 10 | 9 | 19
  United States: Midwest | 4 | 5 | 9
  United States: Southwest | 3 | 5 | 8
  United States: West | 9 | 8 | 17
ATLS Certification [Count of Participants; unit: Participants] — Completion of Advanced Trauma Life Support (ATLS) course, which instructs learners in the American College of Surgeons guidelines for the triage of trauma patients.
  Participants | 31 | 33 | 64
Specialty [Count of Participants; unit: Participants]
  Emergency Medicine | 29 | 30 | 59
  Family Practice | 3 | 1 | 4
  Internal Medicine | 1 | 2 | 3
  Other (e.g. general surgery) | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Signed up for the Intervention That Completed All 3 Coaching Sessions.
Description: A summary of the number of trainees who signed up for coaching sessions and completed all three sessions as assigned.
Time Frame: 3 week intervention period
Population: Board-certified emergency physicians who triage and treat adult patients in the emergency department of either a non-trauma center or a Level III/IV trauma center in the United States.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Participants in the control group who enrolled in the trial.
Arm/Group | Deliberate Practice | Control
Number analyzed (Participants) | 36 | 36
Participants
  Completed 3 coaching sessions | 28 | 0
  Completed 2 coaching sessions | 2 | 0
  Completed 1 coaching session | 0 | 0
  Not assigned to coaching sessions | 6 | 36

2. Secondary Outcome: Under-triage
Description: Proportion of severely injured patients NOT transferred to trauma centers/total number of severely injured patients evaluated during a validated virtual simulation
Time Frame: 3 weeks post-intervention (deliberate practice) or 3 weeks post-enrollment (control)
Population: Physicians who used the virtual simulation. We excluded physicians enrolled in the trial but who did not provide outcome data for analysis.
Measure: Mean (Standard Deviation); unit: proportion of patients under-triaged
Groups:
- Control: Participants in the control group who completed a virtual simulation.
- Deliberate Practice: Participants in the intervention arm who completed a virtual simulation
Arm/Group | Control | Deliberate Practice
Number analyzed (Participants) | 21 | 26
proportion of patients under-triaged | 0.85 (0.36) | 0.51 (0.50)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 13.8, 95% CI 2-sided [2.76 to 69.6]

3. Secondary Outcome: Number of Participants Who Describe Coaching as Acceptable.
Description: Derived from semi-structured interviews conducted by members of the investigative team at the conclusion of the 3 week training period. These interviews will focus on participant perceptions of the acceptability of the intervention.
Time Frame: 2- weeks post intervention
Population: Participants assigned to receive the deliberate practice intervention who completed an interview after the training sessions.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Patients who enrolled in the trial and were randomized to not receive the intervention
Arm/Group | Deliberate Practice | Control
Number analyzed (Participants) | 36 | 36
Participants
  Participants received the intervention and who described it acceptable | 26 | 0
  Participants who received the intervention and did not describe it as acceptable. | 2 | 0
  Participants who received the intervention but did not complete an interview | 2 | 0
  Participants who did not receive the intervention | 6 | 36

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Deliberate Practice | Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

LIMITATIONS AND CAVEATS:
First, we used a passive rather than an active control as the comparator, which may have magnified the effect of the intervention. Second, the differential rate of attrition for completing the virtual simulation in the control and intervention groups could introduce bias, if missingness was not random. Third, we used a simulation to assess behavior, albeit one with evidence of criterion validity, which limited inference about the efficacy of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT05168579/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05168579/SAP_001.pdf
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT05168579/ICF_002.pdf